CLINICAL TRIAL: NCT06481462
Title: Comparison of the Effects of Intrathecal Morphine and Ultrasound-Guided Bilateral Posterior Quadratus Lumborum Block on Postoperative Acute Pain in Cesarean Section: A Prospective, Observational Study
Brief Title: Intrathecal Morphine vs. US-Guided Bilateral Posterior Quadratus Lumborum Block in Cesarean Section
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Doc. Dr, Ondokuz Mayıs University
Other Study IDs: ITMQLB27
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Postoperative Pain
Keywords: Cesarean section; intrathecal morphine; posterior quadratus lumborum block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intrathecal Morphine: A subarachnoid block will be performed by injecting morphine 100 mcg + 12.5 mg hyperbaric bupivacaine + 20 mcg fentanyl.
  Interventions: Procedure: Intrathecal Morphine (ITM)
- Posterior Quadratus Lumborum Block: Patients scheduled for elective cesarean section under spinal anesthesia will receive bilateral ultrasound-guided posterior quadratus lumborum block.
  Interventions: Procedure: Quadratus Lumborum II (QLB-II) Block

INTERVENTIONS:
Procedure: Intrathecal Morphine (ITM) — morphine 100 mcg + 12.5 mg bupivacaine + 20 mcg fentanyl
  Groups: Intrathecal Morphine
Procedure: Quadratus Lumborum II (QLB-II) Block — 12.5 mg bupivacaine + 20 mcg fentanyl bilateral QLB block (posterior tip 2) 25 cc 0.25% bupivacaine
  Groups: Posterior Quadratus Lumborum Block

SUMMARY:
In this study, it was aimed to evaluate the effects of intrathecal morphine and posterior quadratus lumborum block (QLB2) on postoperative acute pain scores and opioid consumption in the first 24 hours after cesarean section.

DETAILED DESCRIPTION:
Postoperative acute pain following a cesarean section is sharp, well-localized, and highly intense. An ideal pain management approach after a cesarean section should provide high-quality analgesia with minimal side effects and facilitate the mother's rapid return to daily activities. Different options for pain control include central blocks, peripheral blocks, and systemic medications.

Intrathecal morphine (ITM) administration is a widely used approach for post-cesarean pain management both globally and in our clinic. However, it can reduce patient satisfaction due to side effects such as nausea, vomiting, and itching. On the other hand, the Quadratus Lumborum Block (QLB), a type of peripheral block, has proven analgesic efficacy in controlling acute postoperative pain following a cesarean section. The aim of this study is to examine and compare the analgesic efficacy of intrathecal morphine (ITM) and Posterior Quadratus Lumborum in the management of acute postoperative pain after a cesarean section.

This study is a single-center, double-blind, prospective observational study.

Patients will be divided into 2 groups.

Group 1: The group receiving intrathecal morphine (ITM)

Group 2: The group receiving Posterior Quadratus Lumborum Block

In elective cesarean section cases under spinal anesthesia, the patient group receiving ITM and posterior QLB will be evaluated for obstetric general well-being during the first 24 hours and at discharge. Total morphine consumption in the first 24 hours, Pain scores (NRS) at rest and during movement, presence of nausea-vomiting and itching, patient satisfaction and any potential side effects will be recorded through follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant for at least 37 weeks
* Aged between 18 and 45
* ASA (American Society of Anesthesiologists) physical status score II
* Patient planned for elective cesarean section under spinal anesthesia
* Patient receiving QLB-II block or intrathecal morphine

Exclusion Criteria:

* ASA score of III or IV.
* Planned cesarean section under general anesthesia.
* Requirement for conversion to general anesthesia after failed spinal anesthesia.
* Contraindication to spinal anesthesia and regional anesthesia techniques.
* BMI greater than 35 kg/m².
* History of opioid use disorder or opioid use for more than 4 weeks.
* Inability to assess pain scores.
* Pregnancies of less than 37 weeks gestation.
* History of allergy to local anesthetics and systemic opioids.
* Patient refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients scheduled for cesarean section at ≥37 weeks of gestation.
Study Population: The study population consisted of pregnant women who were at least 37 weeks gestational age, aged between 18 and 45 years, with an ASA (American Society of Anesthesiologists) physical status score of II, scheduled for elective cesarean section under spinal anesthesia between July 1, 2024, and October 20, 2024, and who received either a posterior quadratus lumborum block (QLB-II) or intrathecal morphine.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured by IV PCA. Patients will be able to request opioids via a PCA device when their NRS score is above 4

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative day 1
  Pain status at rest and while coughing will be assessed by NRS scores at 0, 3, 6, 12, and 24 hours after operation.The NRS is an 11-point numeric scale which ranges from 0 to 10.
Postoperative nausea and vomiting (PONV) scores | Postoperative Day 1
  The severity of postoperative nausea and vomiting (PONV) will be assessed using a descriptive verbal rating scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more, ondansetron 4 mg IV will be administered and will repeat after 8 hours if required. The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
The number of patient required rescue analgesic | Postoperative Day 1
  The number of patient requires rescue analgesic will be recorded at 0, 3, 6, 18, and 24 hours after operation
Postoperative pruritus score | Postoperative Day 1
  Pruritus score: 0 = no pruritus; 1 = sensation of itching, but not scratching, just a rubbing sensation (mild); 2 = sensation of itching and scratching (moderate); 3 = sensation of pruritus, scratching, and requiring treatment (severe).
Patients' satisfaction and quality of pain management | Postoperative Day 1
  Patients' pain management satisfaction and quality will be evaluated using the QoR-11 score. ObsQoR-11 is an 11-item questionnaire that is used to evaluate the recovery of parturient women after elective CS. ObsQoR-11 is evaluated in terms of the degree of post-operative pain, nausea, vomiting, activity, baby care, hygiene,and emotional control. Each item was scored using an 11-point system, with minimum and maximum scores of 0 and 110, respectively. A high score reflects good recovery.
  QoR-11 Turkish Version will be used for assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan DOST, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salama ER. Ultrasound-guided bilateral quadratus lumborum block vs. intrathecal morphine for postoperative analgesia after cesarean section: a randomized controlled trial. Korean J Anesthesiol. 2020 Apr;73(2):121-128. doi: 10.4097/kja.d.18.00269. Epub 2019 Mar 8. PMID 30852882
- [Background] Krohg A, Ullensvang K, Rosseland LA, Langesaeter E, Sauter AR. The Analgesic Effect of Ultrasound-Guided Quadratus Lumborum Block After Cesarean Delivery: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):559-565. doi: 10.1213/ANE.0000000000002648. PMID 29135590
- [Background] Ozkan G, Kara U, Ince ME, Ozdemir O, Ulubay M, Senkal S. Validation of the Turkish version of the Obstetric Quality-of-Recovery score 11 (ObsQoR-11T) after cesarean delivery. Health Qual Life Outcomes. 2022 Nov 28;20(1):155. doi: 10.1186/s12955-022-02073-y. PMID 36443784